CLINICAL TRIAL: NCT04802655
Title: Effect of Exergame Program Structured Via Analytic Hierarchy Process on Trunk Control and Upper Extremity Functionality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmet Emir (Other)
Responsible Party: Sponsor-Investigator, Ahmet Emir, Lecturer, Medipol University
Organization: Medipol University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-10840098-772.02-65173
Record Dates: First submitted 2021-03-15; First posted 2021-03-17 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exergame Group (EG) (Experimental): In addition to routine NDT training, Structured Exergame Program for upper extremity and trunk control will be applied in this group. Xbox one - Kinect supported video games will be selected for video-game based exergame program. The Video games to be included in the Exergame program will be selected by Analytical Hierarchy Process. Program will consist 40 minutes of exergame sessions and 15 sessions total. Sessions will be applied 2 times a week, and It is planned to complete in 8 weeks.
  Interventions: Other: Video-game based exercise - Exergame
- Activity Based Exercise Group (AG) (Active Comparator): In addition to routine NDT training, Goal Directed Activity Based Exercises for upper extremity and trunk will be applied to this group. Program will consist 40 minutes of exergame sessions and 15 sessions total. Sessions will be applied 2 times a week, and It is planned to complete in 8 weeks.
  Interventions: Other: Activity Based Exercise Group (AG)

INTERVENTIONS:
Other: Video-game based exercise - Exergame — Selected Kinect compatible video games from Microsoft Xbox one will be applied in this group. Four video games will be selected for a session (each game will last 10 mins). Video games are active video games which participants have to use their body parts in order to control games.
  Other Names: Microsoft Xbox One Kinect based exergame program
  Arms: Exergame Group (EG)
Other: Activity Based Exercise Group (AG) — Task-oriented exercises to be performed in standing and sitting positions, including upper extremity and trunk, will be applied to the activity-based exercise group in addition to routine NDT training. Examples for activities; stepping and putting stickers on the wall, treading the play dough placed on a step board within one leg stance; reach-grasp activities progressively from sitting to standing, throwing and catching balls on a balance board.
  Other Names: Goal Directed Upper Limb and Postural Control Exercises
  Arms: Activity Based Exercise Group (AG)

SUMMARY:
The aim of the study is to investigate effects of structured exergame program on upper extremity functions and trunk control in children with Cerebral Palsy (SP). A 3 phase randomized controlled trial has planned to conduct. In the first phase, baseline assessments will be completed for all participants who are eligible to participate. After the baseline assessments, randomisation will be completed for Exergame and Activity Based Exercise groups. During this phase suitable video games for exergame program will be selected. Analytical Hierarchy Process (AHP) will be used to collect expert opinion for most effective video games for upper extremity functionality, postural control, GMFCS I-II-III levels. Second phase of the study will be started afterwards. Upon completing second assessments, interventions for both groups will be conducted. Third assessments will be completed after interventions and outcomes will be analyzed for primary results. The third phase of the study planned as follow-up period. All participant will continue their routine NDT trainings and follow-up assessments will be completed after 3 moths of the second assessments. Final results will be analysed for all participants.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with spastic cerebral palsy
* Gross Motor Level should be in between I-III according to Gross Motor Function Classification System (GMFCS)
* Manual ability levels should be in between I-IV according to Manual Abilities Classification System (MACS)
* No Botulinum toxin injections 6 months prior to study

Exclusion Criteria:

* Surgery history related to the musculoskeletal system (upper and lower extremities)
* Having communication problems
* Having secondary cognitive-behavioral problems addition to cerebral palsy (intellectual disability)

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Upper Limb Kinematics - Range of Motion Analysis | 10 minutes
  Upper limb kinematics analysis for range of motion assessments will be conducted via Kinovea 2D motion analysis software. Analysis will be conducted during 1 selected activity which is putting glasses into shelves. Reflective markers will be placed on the lateral side of head, shoulder, elbow and hand. Video recordings will be completed from the affected side of the body laterally. Shoulder, elbow and wrist Range of Motion (ROM) values (in degrees) each pivots will be analyzed afterward.
Upper Limb Kinematics - Angular velocity | 10 minutes
  Upper limb kinematics analysis for angular velocity will be conducted via Kinovea 2D motion analysis software.Analysis will be conducted during 1 selected activity which is putting glasses into shelves. Reflective markers will be placed on the lateral side of head, shoulder, elbow and hand. Video recordings will be completed from the affected side of the body laterally. Shoulder, elbow and wrist angular velocity (mm/s) of each pivots will be analyzed afterward.
Trunk Control Measurement Scale (TCMS) | 15 minutes
  Trunk Control Measurement Scale (TCMS) is a clinical tool to measure trunk control in children with cerebral palsy. TCMS measures the trunk control in two basic components that are static and dynamic sitting balance. Dynamic sitting balance is divided into two parts as selective movement control and dynamic reaching. The static sitting balance part evaluates trunk control during upper and lower limbs' movements in the sitting position. Balance is assessed during flexion, extension, lateral flexion and rotation movements as selective movements of dynamic sitting. Reaching part of dynamic sitting balance evaluates trunk balance during reaching at different planes. The scale consists of 15 items. Each part has 5,7 and 3 items respectively. Total score ranges between0 and 58 and higher scores reflect better control.

SECONDARY OUTCOMES:
Selective Control of Upper Extremity Scale (SCUES) | 15 minutes
  The SCUES is a video-based assessment tool evaluating upper extremity joint levels, including the shoulder, elbow, forearm, wrist, and fingers. The administration of the SCUES required patients to perform specific isolated movement patterns at various levels including: shoulder (abduction/adduction); elbow (flexion/extension); forearm (supination/pronation); wrist (flexion/extension); and fingers/thumb (grasp/release). Presence of mirror movements, movement of additional joints, and any motion less than available ROM are scored for movement at each joint level. Considering these four common manifestations of impaired SMC, motion at each of the five joint levels is scored on a four-point scale as: no SMC (0 point), moderately diminished SMC (1 point), mildly diminished SMC (2 point), and normal SMC (3 point). The total score of the SCUES ranges between 0 and 15 and higher scores indicate better SMC.
Jebsen Taylor Hand Function Test (JTHFT) | 10 minutes
  The JTHFT consists of seven unimanual items that are administered using standardized procedures and verbal instructions and performed first with the nondominant hand and then with the dominant hand. The functional tasks on the JTHFT-IT include (a) writing a 24-letter, third-grade reading difficulty sentence; (b) turning 300-500 (7.62 cm by 12.7 cm) cards in simulated page turning; (c) picking up small common objects (including pennies, paper clips, and bottle caps) and placing them in a container; (d) stacking checkers; (e) simulated feeding; and (f) moving light cans and heavier (1 pound) cans. The subtests are scored by recording with a stopwatch the number of seconds required to complete each task.
Pediatric Evaluation of Disability Inventory - Computer Adaptive Test (PEDI-CAT) | 15 minutes
  The PEDI-CAT is a comprehensive clinical assessment of functional skills acquired throughout infancy, childhood and adolescence up through the age of 20 years. Each of the four PEDI-CAT domains (daily activities, mobility, social/cognitive and responsibility) is independent and can be used separately or in combination with the other domains. Items in three of the domains focus on the child's ability to perform each functional activity in a manner that is effective given their abilities and challenges. The items in the responsibility domain examine the extent to which responsibility management for complex tasks has been shifted from parent to child. Items do not require the child to perform the activity in a standardized manner for scoring.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Emir, Msc, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No